CLINICAL TRIAL: NCT00217204
Title: A Phase II, Randomized, Investigator-Blinded, Parallel-Group, Pilot Study Evaluating the Safety, Palatability and Effectiveness of Four Doses of Pancrelipase Microtablets in the Treatment of Infants and Toddlers With Cystic Fibrosis-Related Pancreatic Insufficiency and Fat Malabsorption
Brief Title: An Effectiveness, Safety, and Palatability Study of Pancrelipase Microtablets in Infants and Toddlers With Cystic Fibrosis and Fat Malabsorption
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR002665
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Cystic Fibrosis; Steatorrhea
Keywords: Cystic fibrosis; Pancreatic insufficiency; Steatorrhea; Fat malabsorption; Pancrelipase
MeSH Terms: conditions — Cystic Fibrosis; Steatorrhea; Exocrine Pancreatic Insufficiency

INTERVENTIONS:
Drug: Pancrelipase microtablets

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of PANCREASE MT (pancrelipase microtablets) to improve steatorrhea (excessive excretion of fat in feces) in infants and toddlers with cystic fibrosis who have pancreatic insufficiency, and to assess whether the consistency of the microtablets is acceptable for swallowing in infants and toddlers

DETAILED DESCRIPTION:
The objective of this randomized, Investigator-blinded, parallel group, multicenter, pilot study is to evaluate the preliminary safety, palatability and effectiveness of pancrelipase microtablets to improve fat absorption. The hypothesis is that PANCREASE MT will provide effective, safe and palatable pancreatic enzyme supplementation to be used for the treatment of fat malabsorption in a cohort of infants with cystic fibrosis-related pancreatic insufficiency. On Day 1 of the study, parents will be instructed to administer 500 units lipase/kg/meal for a full five days. Stool will be collected and analyzed during the last 72 hours of this baseline period. On Day 6 of the study, subjects will be randomly assigned to one of four treatment groups. Parents will be instructed to administer the appropriate dose for a full five days and stool will be collected and analyzed during the last 72 hours of this randomized treatment period. Patients will receive PANCREASE MT 500 units lipase/kg/meal by mouth for a maximum of five doses per day for the first 120 hours. Patients will receive PANCREASE MT 500, 1000, 1500 or 2000 units lipase/kg/meal by mouth, for a maximum of five meals per day for the next 120 hours.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis
* Excessive discharge of fat in feces
* Stable patient requiring pancreatic enzyme therapy

Exclusion Criteria:

* No stable antibiotic therapy for small bowel overgrowth
* No hypersensitivity to pork products
* No use of prokinetics eg, metoclopramide or cisapride within the last 30 days
* No nasogastric feeding tube feeding
* No use of steroids
* No use of concomitant H2 blockers or proton pump inhibitors as concomitant therapy

Ages: 6 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2005-07; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change in coefficient of fecal fat absorption from baseline to end of study period. Palatability. Percent carbon dioxide expired by 13C-mixed triglyceride breath test measuring exogenous lipase activity.

SECONDARY OUTCOMES:
Clinical Global Impression Severity Subscale. Global Change Subscale. Weight gain/loss. Global Assessment effectiveness. Nitrogen excretion/24 hr. Mean dose of pancrease assessed/day & weight. Mean daily calories, fat intake. Coefficient fat absorption

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- See also: An Effectiveness, Safety, and Palatability Study of Pancrelipase Microtablets in Infants and Toddlers With Cystic Fibrosis and Fat Malabsorption — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=907&filename=CR002665_CSR.pdf